CLINICAL TRIAL: NCT03330470
Title: Molecular Mediators of Physical Exercise and Carnosine Induced Effects in Patients With Preclinical and Early Stage Neurodegenerative Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Slovak Academy of Sciences (Other Government)
Collaborators: Comenius University (Other); University Hospital Bratislava (Other); National Cheng Kung University (Other)
Responsible Party: Principal Investigator, Barbara Ukropcová, MD, PhD, Prof. MD, PhD, Slovak Academy of Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 15-0253
Record Dates: First submitted 2017-10-17; First posted 2017-11-06 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Subjective Cognitive Impairment; Mild Cognitive Impairment; Parkinson Disease; Healthy Volunteers
Keywords: Parkinson's disease; exercise training; motor functions; cognitive functions
MeSH Terms: conditions — Cognitive Dysfunction; Parkinson Disease | interventions — Exercise; Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- exercise and carnosine supplementation (Experimental): exercise: participants will be subjected to 4 months of supervised exercise intervention carnosine supplementation: participants will be instructed to take carnosine 2 times daily
  Interventions: Behavioral: exercise; Dietary Supplement: carnosine supplementation
- exercise and supplementation with placebo (Experimental): exercise: participants will be subjected to 4 months of supervised exercise intervention supplementation with placebo: participants will be instructed to take placebo 2 times daily
  Interventions: Behavioral: exercise; Dietary Supplement: supplementation with placebo
- stretching controls and carnosine supplementation (Experimental): stretching controls: participants will be subjected to 4 months of supervised stretching program carnosine supplementation: participants will be instructed to take carnosine 2 times daily
  Interventions: Dietary Supplement: carnosine supplementation; Behavioral: stretching
- stretching controls and supplementation with placebo (Experimental): stretching controls: participants will be subjected to 4 months of supervised stretching program supplementation with placebo: participants will be instructed to take placebo 2 times daily
  Interventions: Behavioral: stretching; Dietary Supplement: supplementation with placebo

INTERVENTIONS:
Behavioral: exercise — participants will be subjected to 4 months supervised exercise intervention
  Arms: exercise and carnosine supplementation; exercise and supplementation with placebo
Dietary Supplement: carnosine supplementation — participants will be instructed to take carnosine 2 times daily
  Arms: exercise and carnosine supplementation; stretching controls and carnosine supplementation
Behavioral: stretching — participants will be subjected to 4 months supervised stretching program
  Arms: stretching controls and carnosine supplementation; stretching controls and supplementation with placebo
Dietary Supplement: supplementation with placebo — participants will be instructed to take placebo 2 times daily
  Arms: exercise and supplementation with placebo; stretching controls and supplementation with placebo

SUMMARY:
The purpose of this study is to investigate the beneficial effects of regular exercise and the impact of food supplement carnosine on cognitive, motoric and metabolic functions as well as on specific biologically active substances in volunteers with subjective (SCI) or mild (MCI) cognitive impairment, as well as in patients in early stages of Parkinson's disease. The investigators assume the immediate intervention-associated health benefit for volunteers.

DETAILED DESCRIPTION:
Standard Operating Procedures for patient recruitment, data collection, data management, data analysis routinely used in Biomedical Research Center, Slovak Academy of Sciences, University Hospital Bratislava and Comenius University, Bratislava will be employed. Gait and balance parameters will be examined and analysed at the Department of Behavioural Neuroscience, Centre of Experimental Medicine, Slovak Academy of Sciences, Bratislava, Slovakia Statistical analysis will be employed to address the primary and secondary objectives, as specified in the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age 55 - 80 years
* Presence of Subjective Cognitive Impairment (SCI), Mild Cognitive Impairment (MCI) or early stage of Parkinson's Disease (Hoehn-Yahr 1st-2nd stage), assessed by experienced neurologist

Exclusion Criteria:

* Serious systemic cardiovascular, hepatic, renal disease, cancer
* Lack of compliance

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
glucose tolerance | up to 36 months
  changes in glucose tolerance will be determined with oral glucose tolerance test (2h glucose, mmol/l)
learning/working memory | up to 36 months
  exercise related changes in learning/working memory will be determined with the aid of Addenbrook's cognitive test (maximum test score 100)
Balance parameter (Berg Balance Scale) | up to 36 months
  Exercise related changes in ballance will be examined with the Berg Balance Scale test (max score 56)

SECONDARY OUTCOMES:
habitual physical activity | up to 36 months
  Habitual physical activity will be determined with accelerometers
physical fitness | up to 36 months
  Submaximal aerobic capacity will be determined with one mile (Rockport) walk test
Gait parameters (Walking speed) | 24 months
  Walking (gait) speed will be evaluated in a subset of PD individuals with the Azure Kinect depth camera (once the technology for gait analysis will be available to the study investigators). An average walking velocity will be computed as total distance divided by time of the test (m·s-¹); measured using Microsoft Kinect for Azure
Gait parameter (Stance time) | 24 months
  Stance time will be evaluated in a subset of PD individuals, (once the technology for gait analysis will be available to the study investigators). Stance time - duration within the gait cycle when the measured leg is in contact with the ground. Measured using Microsoft Kinect for Azure as the time from when ankle joint speed in the anterior-posterior direction drops below 10% of its peak to reaching 10% in the next gait cycle, unit measure (s)
Gait parameter (step length) | 24 months
  Step length - linear distance in the anterior-posterior direction between consecutive heel strikes of opposite feet (m); measured using Microsoft Kinect for Azure as the peak distance between left and right ankle points. In a subpopulation of PD patients after (Azure Kinect) technology is available.
Postural parameter (magnitude of CoP displacement) | 24 months
  Magnitude of centre of pressure (CoP) displacement - exercise-related changes in CoP magnitude in both anterior-posterior and medial-lateral directions reflecting the whole body sway will be determined with the aid of force platform (mm)
Postural parameter (Velocity CoP displacement) | 24 months
  Velocity of centre of pressure (CoP) displacement - exercise-related changes in CoP velocity in both anterior-posterior and medial-lateral directions reflecting the whole body sway will be determined with the aid of force platform (mm/s)
Postural Sway Area | 24 months
  Postural sway area - exercise-related changes in the overall centre of pressure (CoP) displacement over a period of time computed as the area enclosed by the CoP path per unit of time will be determined with the aid of force platform (mm-2.s-1)
Postural sway path length | 24 months
  Postural sway path length - exercise-related changes in the overall centre of pressure (CoP) displacement computed as the total distance the CoP travels will be determined with the aid of force platform (mm)
Postural sway frequency | 24 months
  Postural sway frequency - exercise-related changes in the rate of the centre of pressure (CoP) oscillations in both anterior-posterior and medial-lateral directions will be determined with the aid of force platform using time-domain and frequency domain analyses (Hz)
Acceleration of upper and lower trunk | 24 months
  Acceleration of upper and lower trunk - exercise-related changes in acceleration of upper and lower trunk in both anterior-posterior and medial-lateral directions reflecting the upper body sway will be determined with the aid of inertial sensors with inbuilt 3D accelerometers (m-2)
Upper and lower trunk sway area | 24 months
  Upper and lower trunk sway area - exercise-related changes in the overall acceleration of upper and lower trunk over a period of time computed as the area enclosed by the acceleration path per unit of time will be determined with the aid of inertial sensors with inbuilt 3D accelerometers (m-2.s-5)
Upper and lower trunk sway path | 24 months
  Upper and lower trunk sway path - exercise-related changes in the overall acceleration of upper and lower trunk computed as the total length of the acceleration path will be determined with the aid of inertial sensors with inbuilt 3D accelerometers (m.s-2)
Upper and lower trunk sway frequency | 24 months
  Upper and lower trunk sway frequency - exercise-related changes in the rate of upper and lower trunk acceleration in both anterior-posterior and medial-lateral directions will be determined with the aid of inertial sensors with inbuilt 3D accelerometers using time-domain and frequency domain analyses (Hz)
Upper and lower trunk sway jerkiness | 24 months
  Upper and lower trunk sway jerkiness - exercise-related changes in the jerk of upper and lower trunk computed as a time derivative of upper and lower trunk acceleration will be determined with the aid of inertial sensors with inbuilt 3D accelerometers (m-2.s-5)
Angular velocity of upper and lower trunk | 24 months
  Angular velocity of upper and lower trunk - exercise-related changes in angular velocity of upper and lower trunk in both anterior-posterior and medial-lateral directions will be determined with the aid of inertial sensors with inbuilt 3D gyroscopes (rad.s-1)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Turčáni, Prof., MD, PhD, Principal Investigator — University Hospital Bratislava, Comenius University, Bratislava,; Peter Valkovič, Prof., MD, PhD, Principal Investigator — University Hospital Bratislava, Comenius University, Bratislava,; Barbara Ukropcová, Assoc. Prof., MD, PhD, Principal Investigator — Biomedical Research Center, Slovak Academy of Sciences,; Jozef Ukropec, DrSc, PhD, Principal Investigator — Biomedical Research Center, Slovak Academy of Sciences,
Locations (3):
- Slovakia (2):
  - University Hospital Bratislava, Comenius University, Bratislava
  - Biomedical Research Center, Slovak Academy of Sciences, Bratislava
- Laboratory of Cognitive Neurophysiology, Institute of Physical Education, Health & Leisure Studies, National Cheng Kung University, Tainan, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No